CLINICAL TRIAL: NCT01501045
Title: The Effect of Transmagnetic Stimulation on Descending Pain Modulation
Brief Title: Effect of Transmagnetic Stimulation on Conditioned Pain Modulation (CPM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, d_yarnitsky, head of Neurology Department, Rambam Health Care Campus
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: TMS-001
Record Dates: First submitted 2011-12-12; First posted 2011-12-29 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Headache; Migraine
Keywords: TMS; CPM; headache; migraine; EEG; psychophysics
MeSH Terms: conditions — Headache; Migraine Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- healthy subjects (Experimental): healthy subjects
  Interventions: Device: TMS system MagPro x100, Tonica Elektronik A/S, Denmark
- pain patients (Experimental): Migraine and muscle headache patients
  Interventions: Device: TMS system MagPro x100, Tonica Elektronik A/S, Denmark

INTERVENTIONS:
Device: TMS system MagPro x100, Tonica Elektronik A/S, Denmark — repeated TMS (rTMS)
  Other Names: Transcranial Magnetic Stimulator
  Arms: healthy subjects
Device: TMS system MagPro x100, Tonica Elektronik A/S, Denmark — repeated TMS
  Other Names: Transcranial Magnetic Stimulator
  Arms: pain patients

SUMMARY:
While some indications of the neural circuits involved in the Conditioned Pain Modulation (CPM) process are now available, there is still need to clarify what parts of the brain are essential for this process, whether the spino-brainstem loop is largely sufficient to explain CPM or whether other cerebral and spinal regions such as frontal, somatosensory and other cortical regions contribute substantially. Whereas mere observation of correlation between these circuits while activated by brain imaging is still of considerable interest, direct experimental manipulations by repetitive transcranial magnetic stimulation (rTMS) could even establish insights into causal relationships.

DETAILED DESCRIPTION:
rTMS of different intensities, frequencies and location will be applied during CPM to evaluate the central mechanisms of pain modulation, their location and role in pain reduction through enhancement or suppression of activity in the relevant brain regions. In other words, cortical regions that may be implicated in CPM will be determined by augmenting or interrupting their activity via rTMSapplied to the areas under investigation. The regions will be the pain network sites, which are assumed to control the top-down influence on CPM and are superficial enough to be stimulated by the magnetic coil. These include primarily DLPFC (dorsolateral prefrontal cortex) and OFC (orbitofrontal cortex), with possible later addition of other relevant sites such as ACC (anterior cortex cinguli), insula and somatosensory cortices, etc. Since rTMS may be administered in a manner that either reduces or enhances the excitability of the stimulated cortical region, it should be possible to clarify the inhibitory or excitatory role of these regions in the CPM process. In summary, the planned studies should allow for identifying the cortical regions of the descending pain system, which are critical as starting points for the top-down modulation of CPM.

ELIGIBILITY:
Inclusion Criteria:

* age 18-70
* males and females
* right handed

Exclusion Criteria:

* metal in brain/skull
* cardiac pacemaker
* cohlear implants
* history of head trauma
* history of epilepsy or seizures
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
Pain scores as measured by pain numerical scale (NPS) | 1 week
  TMS directed to pain inhibitory cortical areas will evoke pain reduction
Amplitude of pain-evoked potentials | 1 week
  Change in pain evoked potentials will be assessed before and after the TMS

SECONDARY OUTCOMES:
conditioned pain modulation (CPM) | 1 week
  Change in the efficiency of CPM will be assessed in response to TMS

CONTACTS AND LOCATIONS:
Overall Officials: David Yarnitsky, professor, Principal Investigator — Rambam Health Care Campus
Locations (1):
- The lab of clinical neurophysiology, the faculty of medicine, Technion and Rambam Medical Center, Haifa, Israel